CLINICAL TRIAL: NCT02337894
Title: Effects of Nutritional Supplementation With Amino Acids on Liver Lipid Content, Whole-body Protein Turnover, and Body Composition in Obese Pre-pubertal Children
Brief Title: Effects of Amino Acid Supplementation on Liver Lipid Content and Protein Metabolism in Obese Children
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not funded
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 203454
Record Dates: First submitted 2014-12-02; First posted 2015-01-14 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Liver Steatosis; Insulin Resistance; Whole Body Protein Metabolism; Body Composition, Beneficial
Keywords: Protein kinetics; liver steatosis
MeSH Terms: conditions — Fatty Liver; Insulin Resistance; Glucocorticoid Receptor Deficiency | interventions — Amino Acids, Essential; Arginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Essential amino acids plus arginine (Experimental): Children randomized to the intervention group will receive a supplement containing essential amino acids plus arginine in the form of a drink which they will have to take for 8 weeks. Measurement of liver lipid content, hepatic apoptosis, plasma lipids, apolipoprotein B-100 levels, hepatic fatty oxidation, whole body insulin sensitivity, body composition and whole body protein turnover will be compared with the the placebo group, and before and after the intervention.
  Interventions: Dietary Supplement: Essential amino acids plus arginine
- Control drink (Placebo Comparator): The control drinks will be indistinguishable from the intervention drinks in taste and volume, but will contain placebo rather than essential amino acids plus arginine.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Essential amino acids plus arginine — Flavored drink containing essential amino acids plus arginine.
  Arms: Essential amino acids plus arginine
Dietary Supplement: Placebo — Flavored drink without essential amino acids plus arginine.
  Arms: Control drink

SUMMARY:
The purpose of this study is to assess the effect of an eight-week dietary supplementation with essential amino acids plus arginine on liver and plasma lipid content, whole-body fat oxidation, whole-body insulin sensitivity, whole body protein metabolism, and body composition in obese pre-pubertal children.

DETAILED DESCRIPTION:
Up to thirty-two obese pre-pubertal children will be recruited for this study. Up to sixteen will be boys and up to sixteen will be girls. The study will be a double-blinded, placebo-controlled trial using a randomized, but counter-balanced design. This will ensure equal numbers in the two groups that the children are randomized to, for each sex. The control group will receive placebo and the intervention group will receive essential amino acids plus arginine. The supplements (essential amino acids plus arginine, and placebo) will be given in the form of a drink twice a day for a total of 8 weeks. Both the participants and the investigators will be blinded to group assignment.

The primary endpoints of this study are to assess the effect of essential amino acids (EAA) plus arginine supplementation on lipid and protein metabolism. For this, liver lipid content, hepatic apoptosis, plasma lipids, apolipoprotein B-100 (apo B-100) levels, hepatic fatty oxidation, whole body insulin sensitivity, body composition and whole body protein turnover. will be compared between the intervention and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy boy or girl
* Age 7-10 years of age and Tanner stage no greater than stage 1
* BMI ≥ 95th percentile
* Not participating for more than 1 hour/week in a regular physical activity program

Exclusion Criteria:

* Tanner stage greater than stage 1
* Having known chronic illnesses/disorders that may independently affect study outcome measures: type 2 or type 1 diabetes mellitus, neurologic (e.g. epilepsy), neurobehavioral (e.g. Attention deficit disorder and hyperactivity, ADHD) endocrine, hepatic, autoimmune, cardiac and renal disorders. Also, chronic lung disorders except well controlled asthma that does not require permanent use of inhaled/oral steroids
* Taking permanent medications: thyroid hormone replacement therapy, inhaled/oral steroids, insulin, metformin, anabolic drugs (growth hormone replacement therapy and oxandrolone) anti-lipid medication, blood pressure medication, ADHD medication (methylphenidate, amphetamines, atomoxetine)

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-01-30 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Serum levels of markers of lipid metabolism before and after 8 weeks of supplementation with essential amino acids plus arginine vs placebo. | Baseline and 8 weeks
  Change in serum levels of triglycerides, cholesterol, very low density lipoprotein (VLDL), low density lipoprotein (LDL), beta-hydroxybutyrate, Apo-lipoprotein B and plasma cytokeratin 18 will be assessed after 8 weeks of essential amino acids plus arginine vs placebo.
Liver lipid content before and after 8 weeks of supplementation with essential amino acids plus arginine vs placebo. | Baseline and 8 weeks
  Nuclear Magnetic Resonance Spectroscopy will be used to assess changes in liver lipid content following an 8-week supplementation period with essential amino acids plus arginine vs. placebo.
Whole body protein turnover before and after 8 weeks of supplementation with essential amino acids plus arginine vs. placebo. | Baseline and 8 weeks
  Change in whole body protein metabolism (synthesis and breakdown) following 8 weeks of essential amino acids plus arginine vs placebo. This outcome will be assessed using a stable isotope of an amino acid (15N-alanine).
Body composition before and after 8 weeks of supplementation with essential amino acids plus arginine vs. placebo. | Baseline and 8 weeks
  Changes in body composition (fat free mass and fat mass) will be assessed using Dual-Energy X-ray Absorptiometry. Measurements will be carried out at baseline and following 8 weeks of supplementation with essential amino acids plus arginine vs. placebo.

SECONDARY OUTCOMES:
HOMA-IR index before and after 8 weeks of supplementation with essential amino acids plus arginine vs placebo. | Baseline and 8 weeks
  Fasting glucose and insulin levels will be used to assess changes in the HOMA-IR index after 8 weeks of supplementation with essential amino acids plus arginine vs. placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Diaz, MD, Principal Investigator — University of Arkansas; Elisabet Borsheim, Ph.D, Study Director — University of Arkansas

REFERENCES:
- [Background] Borsheim E, Bui QU, Tissier S, Cree MG, Ronsen O, Morio B, Ferrando AA, Kobayashi H, Newcomer BR, Wolfe RR. Amino acid supplementation decreases plasma and liver triacylglycerols in elderly. Nutrition. 2009 Mar;25(3):281-8. doi: 10.1016/j.nut.2008.09.001. Epub 2008 Nov 28. PMID 19041223
- [Background] Borsheim E, Bui QU, Tissier S, Kobayashi H, Ferrando AA, Wolfe RR. Effect of amino acid supplementation on muscle mass, strength and physical function in elderly. Clin Nutr. 2008 Apr;27(2):189-95. doi: 10.1016/j.clnu.2008.01.001. Epub 2008 Mar 4. PMID 18294740
- [Background] van Vught AJ, Heitmann BL, Nieuwenhuizen AG, Veldhorst MA, Brummer RJ, Westerterp-Plantenga MS. Association between dietary protein and change in body composition among children (EYHS). Clin Nutr. 2009 Dec;28(6):684-8. doi: 10.1016/j.clnu.2009.05.001. Epub 2009 Jun 12. PMID 19524336